CLINICAL TRIAL: NCT03959423
Title: Safety Evaluation of the Advanced Hybrid Closed Loop (AHCL) System in Type 1 Adult and Pediatric Subjects
Brief Title: Safety Evaluation of the Advanced Hybrid Closed Loop (AHCL) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP321
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects 7-75 years of age (Experimental): Subjects who have been diagnosed with type 1 diabetes
  Interventions: Device: AHCL insulin pump system

INTERVENTIONS:
Device: AHCL insulin pump system — 670G 4.0 system with GS3; 780G system with G4S (continued access phase);

SUMMARY:
This study is a Safety Evaluation of the Advanced Hybrid Closed Loop (AHCL) System in Type 1 Adult and Pediatric Subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety of the Advanced Hybrid Closed Loop system (AHCL) in type 1 diabetes adult and pediatric subjects in a home setting. The main objective in conducting this research is to collect data from patients who use the AHCL system at home, at work, at school and everywhere else. Subjects will use 670G 4.0 system with Guardian Sensor 3 (GS3) during study period, and will be allowed to participate in continued access phase, and use 670G 4.0 system with GS3 and 780G system with Guardian 4 Sensor (G4S).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 7-75 years at time of Screening
2. Subjects 14-75 years of age: A clinical diagnosis of type 1 diabetes for 2 years or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Subjects 7-13 years of age: A clinical diagnosis of type 1 diabetes for 1 year or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis Study-specific inclusion criteria
4. Subject is willing to perform ≥ 4 finger stick blood glucose measurements daily
5. Subject is willing to perform required sensor calibrations
6. Subject is willing to wear the system continuously throughout the study
7. Subject must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units
8. Subject has a Glycosylated hemoglobin (HbA1c) less than 10% (as processed by Central Lab) at time of Screening visit Note: All HbA1c blood specimens will be sent to and tested by a NGSP certified Central Laboratory. HbA1c testing must follow National Glycohemoglobin Standardization Program (NGSP) standards.
9. Subject has TSH in the normal range OR if the TSH is out of normal reference range the Free T3 is below or within the lab's reference range and Free T4 is within the normal reference range.
10. Pump therapy for greater than 6 months prior to screening (with or without CGM experience)
11. Subject must have a companion or caregiver available at night for the duration of the study period who resides (or will live) in in the same building (or home). A companion or caregiver should also be available during exercise challenges in the same building, home or location (if not at home). This requirement may be verified by subject report at screening visit.
12. Subject willing to upload data from the study pump, must have Internet access and a computer system that meets the requirements for uploading the study pump
13. If subject has celiac disease, it has been adequately treated as determined by the investigator
14. Subject is willing to take one of the following insulins and can financially support the use of either of the 2 insulin preparations throughout the course of the study (i.e. co-payments for insulin with insurance or able to pay full amount)

    * Humalog™* (insulin lispro injection)
    * NovoLog™* (insulin aspart)
15. Subjects with history of cardiovascular event 1 year or more from the time of screening must have an EKG within 6 months prior to screening or during screening. If subject has an abnormal EKG, participation is allowed if there is clearance from a cardiologist
16. Subjects with the 3 or more cardiovascular risk factors listed below must have an EKG within 6 months prior to screening or during screening. If subject has an abnormal EKG, participation is allowed if there is clearance from a cardiologist

    a. Cardiovascular risk factors include:
    * Age >35 years
    * Type 1 diabetes of >15 years' duration
    * Presence of any additional risk factor for coronary artery disease
    * Presence of microvascular disease (proliferative retinopathy or nephropathy, including microalbuminuria)
    * Presence of peripheral vascular disease
    * Presence of autonomic neuropathy
17. Subjects with history of cardiovascular event 1 year or more from the time of screening must have a stress test within 6 months prior to screening or during run in period. If subject fails stress test, participation is allowed if there is clearance from a cardiologist

Exclusion Criteria:

1. Subject has a history of 1 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to Screening:

   1. Medical assistance (i.e. Paramedics, Emergency Room (ER) or Hospitalization)
   2. Coma
   3. Seizures
2. Subject has been hospitalized or has visited the ER in the 6 months prior to Screening resulting in a primary diagnosis of uncontrolled diabetes
3. Subject has had Diabetic Ketoacidosis (DKA) in the 6 months prior to Screening.
4. Subject has Hypoglycemia Unawareness, as measured by the Gold questionnaire (Gold, MacLeod et al. 1994) at Screening
5. Subject is unable to tolerate tape adhesive in the area of sensor placement
6. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection)
7. Women of child-bearing potential who have a positive pregnancy test at Screening or plan to become pregnant during the course of the study
8. Females who are sexually active and able to conceive will be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study as determined by investigator.
9. Subject has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
10. Subject is being treated for hyperthyroidism at time of Screening
11. Subject has a diagnosis of adrenal insufficiency
12. Subject has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of Screening, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study
13. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
14. Subject is currently abusing illicit drugs
15. Subject is currently abusing marijuana
16. Subject is currently abusing prescription drugs
17. Subject is currently abusing alcohol
18. Subject is using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of Screening
19. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
20. Subject has elective surgery planned that requires general anesthesia during the course of the study
21. Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of Screening
22. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
23. Subject diagnosed with current eating disorder such as anorexia or bulimia
24. Subject has been diagnosed with chronic kidney disease that results in chronic anemia
25. Subject has a hematocrit that is below the normal reference range of lab used.
26. Subject is on dialysis
27. Subject has serum creatinine of >2 mg/dL.
28. Research staff involved with the study.

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Arkansas Diabetes and Endocrinology Center, Little Rock, Arkansas
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - SoCal Diabetes, Torrance, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center - Adults, Aurora, Colorado
  - Barbara Davis Center - Pediatric, Aurora, Colorado
  - Yale Diabetes Research Program, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Southeastern Endocrine, Roswell, Georgia
  - Rocky Mountain Diabetes Center, Idaho Falls, Idaho
  - International Diabetes Center, Minneapolis, Minnesota
  - AM Diabetes & Endocrinology Center, Bartlett, Tennessee
  - Texas Endocrinology, Austin, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - Rainier Clinical Research, Renton, Washington
  - Seattle Children's Hospital and Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pihoker C, Shulman DI, Forlenza GP, Kaiserman KB, Sherr JL, Thrasher JR, Buckingham BA, Kipnes MS, Bode BW, Carlson AL, Lee SW, Latif K, Liljenquist DR, Slover RH, Dai Z, Niu F, Shin J, Jonkers RAM, Roy A, Grosman B, Vella M, Cordero TL, McVean J, Rhinehart AS, Vigersky RA; MiniMed AHCL Study Group. Safety and Glycemic Outcomes During the MiniMedTM Advanced Hybrid Closed-Loop System Pivotal Trial in Children and Adolescents with Type 1 Diabetes. Diabetes Technol Ther. 2023 Nov;25(11):755-764. doi: 10.1089/dia.2023.0255. Epub 2023 Oct 25. PMID 37782145
- [Derived] Cordero TL, Dai Z, Arrieta A, Niu F, Vella M, Shin J, Rhinehart AS, McVean J, Lee SW, Slover RH, Forlenza GP, Shulman DI, Pop-Busui R, Thrasher JR, Kipnes MS, Christiansen MP, Buckingham BA, Pihoker C, Sherr JL, Kaiserman KB, Vigersky RA. Glycemic Outcomes During Early Use of the MiniMed 780G Advanced Hybrid Closed-Loop System with Guardian 4 Sensor. Diabetes Technol Ther. 2023 Sep;25(9):652-658. doi: 10.1089/dia.2023.0123. Epub 2023 Jun 16. PMID 37252734
- [Derived] Carlson AL, Sherr JL, Shulman DI, Garg SK, Pop-Busui R, Bode BW, Lilenquist DR, Brazg RL, Kaiserman KB, Kipnes MS, Thrasher JR, Reed JHC, Slover RH, Philis-Tsimikas A, Christiansen M, Grosman B, Roy A, Vella M, Jonkers RAM, Chen X, Shin J, Cordero TL, Lee SW, Rhinehart AS, Vigersky RA. Safety and Glycemic Outcomes During the MiniMed Advanced Hybrid Closed-Loop System Pivotal Trial in Adolescents and Adults with Type 1 Diabetes. Diabetes Technol Ther. 2022 Mar;24(3):178-189. doi: 10.1089/dia.2021.0319. Epub 2021 Nov 16. PMID 34694909

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 329 subjects (179 with age 7-17 and 150 with age 18-75) enrolled at the beginning, with 25 (10 with age 7-17 and 15 with age 18-75) screen failure, 15 subjects (8 with age 7-17 and 7 with age 18-75) early withdrawn, and 1 subject (age 7-17) who never used AHCL, 288 subjects (160 with age 7-17 and 128 with age 18-75) were left as the Intention to Treat Population and started the study. After completing the study, 207 (130 with age 7-17 and 77 with age 18-75) entered the Continued Access Period
Groups:
- Subjects 7-17 Years of Age: Subjects 7-17 years of age wearing Advanced Hybrid Closed Loop pump system and using AHCL during Study Period
- Subjects 18-75 Years of Age: Subjects 18-75 years of age wearing Advanced Hybrid Closed Loop pump system and using AHCL during Study Period
Period: Overall Study
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-75 Years of Age
Started | 160 | 128
Completed | 151 | 124
Not Completed | 9 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 6 | 0

BASELINE CHARACTERISTICS:
Population: Intention to Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-75 Years of Age | Total
Number analyzed (Participants) | 160 | 128 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (2.5) | 43.5 (15.2) | 25.6 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 69 | 152
  Male | 77 | 59 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 148 | 120 | 268
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 1 | 5
  White | 144 | 123 | 267
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 4 | 2 | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 19.7 (3.5) | 28.4 (5.6) | 23.6 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: The overall mean difference of the change in HbA1c from baseline to end of 3-month Study Period.
Time Frame: Baseline to End of 3-Month Study Period
Population: Intention to Treat Population with available data. Twenty-four subjects aged 7-17 and one subject aged 18-75 did not collect A1C at the end of the study period, so 136 subjects aged 7-17 and 127 subjects aged 18-75 were analyzed at end of study period and the change from baseline to end of study period.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-75 Years of Age
Number analyzed (Participants) | 160 | 128
percentage
  Baseline | 7.9 (0.9) | 7.4 (0.8)
  End of Study: number analyzed (Participants) | 136 | 127
  End of Study | 7.4 (0.7) | 6.9 (0.5)
  Change from Baseline to End of Study: number analyzed (Participants) | 136 | 127
  Change from Baseline to End of Study | -0.5 (0.7) | -0.5 (0.6)

2. Primary Outcome: Change in Percentage of Euglycemia
Description: The overall mean change in % of time in euglycemia (70-180 mg/dL) from baseline to end of 3-month Study Period will be estimated.
Time Frame: Baseline to End of 3-Month Study Period
Population: Intention to Treat Population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-75 Years of Age
Number analyzed (Participants) | 160 | 128
percentage
  Baseline | 59.4 (11.8) | 70.5 (9.8)
  3 Months Study Period | 70.3 (6.5) | 75.0 (7.2)
  Change from Baseline to 3 Months Study Period | 11.0 (9.1) | 4.6 (5.9)

3. Secondary Outcome: Number of Severe Hypoglycemic Event
Description: Number of severe hypoglycemic events occurred during 3-month Study Period
Time Frame: 3-month Study Period
Population: Intention to Treat Population
Measure: Number; unit: Events
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-75 Years of Age
Number analyzed (Participants) | 160 | 128
Events | 0 | 0

4. Secondary Outcome: Number of Diabetic Ketoacidosis (DKA) Event
Description: Number of Diabetic Ketoacidosis (DKA) event occurred during 3-month Study Period
Time Frame: 3-month Study Period
Population: Intention to Treat Population
Measure: Number; unit: Events
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-75 Years of Age
Number analyzed (Participants) | 160 | 128
Events | 0 | 0

5. Secondary Outcome: Change in Percent of Time in Hypoglycemic Range (<70 mg/dL)
Description: The overall mean change in % of time in hypoglycemic range (<70 mg/dL) from baseline to end of 3-month Study Period will be estimated.
Time Frame: Baseline to End of 3-Month Study Period
Population: Intention to Treat Population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-75 Years of Age
Number analyzed (Participants) | 160 | 128
percentage
  Baseline | 2.7 (2.0) | 3.4 (3.0)
  3 Months Study Period | 2.7 (1.6) | 2.3 (1.7)
  Change from Baseline to 3 Months Study Period | -0.0 (1.7) | -1.0 (2.2)

ADVERSE EVENTS:
Time Frame: 3-month Study Period and 42-month Continued Access Phase
Groups:
- Subjects 7-17 Years of Age Study Period: Subjects 7-17 years of age wearing Advanced Hybrid Closed Loop pump system and using AHCL during Study Period
- Subjects 18-75 Years of Age Study Period: Subjects 18-75 years of age wearing Advanced Hybrid Closed Loop pump system and using AHCL during Study Period
- Subjects 7-17 Years of Age Continued Access Phase: Subjects 7-17 years of age wearing Advanced Hybrid Closed Loop pump system and using AHCL during Continued Access Phase
- Subjects 18-75 Years of Age Continued Access Phase: Subjects 18-75 years of age wearing Advanced Hybrid Closed Loop pump system and using AHCL during Continued Access Phase
Arm/Group | Subjects 7-17 Years of Age Study Period | Subjects 18-75 Years of Age Study Period | Subjects 7-17 Years of Age Continued Access Phase | Subjects 18-75 Years of Age Continued Access Phase
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/128 | 0/130 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/160 | 3/128 | 3/130 | 8/77
Other Adverse Events (participants affected / at risk) | 72/160 | 44/128 | 99/130 | 64/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects 7-17 Years of Age Study Period (N=160) | Subjects 18-75 Years of Age Study Period (N=128) | Subjects 7-17 Years of Age Continued Access Phase (N=130) | Subjects 18-75 Years of Age Continued Access Phase (N=77)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects 7-17 Years of Age Study Period (N=160) | Subjects 18-75 Years of Age Study Period (N=128) | Subjects 7-17 Years of Age Continued Access Phase (N=130) | Subjects 18-75 Years of Age Continued Access Phase (N=77)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Growth hormone deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Primary hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-proliferative retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Malpositioned teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site bruise (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Medical device site dermatitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site erosion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Medical device site haemorrhage (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Medical device site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site rash (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 35 (42) | 33 (38)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (6) | 1 (1) | 10 (11) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 3 (4) | 4 (4)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 7 (7) | 0 (0) | 7 (7) | 4 (4)
Infusion site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (5) | 2 (5) | 3 (3)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 4 (6) | 4 (4)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pitted keratolysis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 4 (4) | 6 (7)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 6 (6) | 20 (28) | 13 (14)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 8 (9) | 2 (5) | 11 (13) | 3 (7)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 7 (9) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypobarism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Incision site vesicles (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 6 (6) | 4 (4)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Poisoning deliberate (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord injury sacral (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Colonoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary scan (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acetonaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (9) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 29 (31) | 2 (2) | 47 (114) | 13 (18)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (5)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Short stature (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Notalgia paraesthetica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Device issue (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tic (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prepuce redundant (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ex-tobacco user (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel decompression (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon sheath incision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03959423/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT03959423/SAP_001.pdf